CLINICAL TRIAL: NCT02296515
Title: Intrathecal Pump Refill: Reservoir Fill Port Identification by Palpation Versus Ultrasound,a Mono-centre Prospective Comparison Study in Patients Undergoing Regular Intrathecal Pump Refill
Brief Title: Intrathecal Pump Refill Undergoing Regular Intrathecal Pump Refill
Status: Completed | Type: Observational
Sponsor: Dr med. Paolo Maino Viceprimario Anestesiologia (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Sponsor-Investigator, Dr med. Paolo Maino Viceprimario Anestesiologia, Dr. med deputy Head of the Anesthisiology, Ospedale Regionale di Lugano
Organization: Ospedale Regionale di Lugano (Other)
Other Study IDs: NSI_TD_001
Record Dates: First submitted 2014-11-05; First posted 2014-11-20 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intrathecal pump refill: — Two different experienced clinicians will perform one time the blind technique andTwo different experienced clinicians will perform one time the blind technique andtwo times the ultrasound-guided technique on all patients.

SUMMARY:
Reservoir fill port identification by palpation versus ultrasound,a mono-centre prospective comparison study in patients undergoing regular intrathecal pump refill

DETAILED DESCRIPTION:
Intrathecal drug therapy with implantable intrathecal pumps is being utilized increasingly for the treatment of chronic refractory pain and spasticity. However, performing the regular refill procedures of the pumps with the commonly performed "blind" technique caries the potential risk of medication injection into the subcutaneous tissue, which can lead to an overdose.

Objective: The primary purpose of this study is to assess the accuracy of the ultrasound-guided technique for the refill procedure compared to the blind technique in subjects undergoing regular refills of their intrathecal pumps for the treatment of chronic non-malignant pain or spasticity.

Study design: Mono-center prospective efficacy and reliability study comparing two approaches to enter the fill port. Study population: The investigators will include patients with an intrathecal pump for the treatment of chronic non-malignant pain or spasticity, undergoing regular refills of their intrathecal pumps at our Centro Terapia del Dolore at the Ospedale Italiano a Viganello(EOC, Switzerland). Intervention: Two different experienced clinicians will perform one time the blind technique and two times the ultrasound-guided technique on all patients.sample size calculations can be performed. The sample size i.e. n=25 patients in NSI-TD-001 Protocol v. 1.0 Final: August 4th, 2014 Confidential Page 31 of 40 total assessed 6 six times is therefore based on practical grounds related feasibility to duration of inclusion (i.e. one year). This would imply 50 paired assessments for both fill port accuracy assessment and intra-rater reliability. The investigators believe based on clinical experience that this number would suffice to detect a difference between methods. Likewise, although no formal power calculation are available for ICC based reliability assessment, as a rule of thumb 50 paired assessments are usually considered adequate to evaluate intra-rater liability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of enrollment;
* The patients are treated for chronic non-malignant pain or spasticity with an intrathecal
* programmable infusion pump and undergo regular refills of their pumps in our clinic.
* Able to provide adequate given written, informed consent to participate in this study.

Exclusion Criteria:

* patient refusal to participate or provide informed consent standard exclusions; pregnancy, lactation, treatment with other investigational products.
* other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction,
* cardiovascular disease).
* infection at the puncture site -participation in another study.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with an intrathecal pump for the treatment of chronic non-malignant pain or spasticity, undergoing regular refills of their intrathecal pumps at our Centro Terapia del Dolore at the Ospedale Italiano a Viganello(EOC, Switzerland).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the number of attempts to enter the reservoir fill port. | 1 YearThe sample size i.e. n=25 patients in total
  The time to perform refill, and patient comfort associated with both procedures will be registered in order to assess user friendliness of both procedures.

SECONDARY OUTCOMES:
the number of skin puncturs | 1 YearYearThe sample size i.e. n=25 patients in total
reliability of the US guided procedure | 1 YearYearThe sample size i.e. n=25 patients
- time to perform refill (usability) | 1 YearYearThe sample size i.e. n=25 patients
patient discomfort | 1 YearYearThe sample size i.e. n=25 patients
- determine if BMI has an impact on the accuracy (the number of attempts) of the two techniques | 1 YearYearThe sample size i.e. n=25 patients

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Maino, Principal Investigator — Ospedale Regionale di Lugano
Locations (1):
- Centro del Dolore, Neurocentro, Opedale Regionale di Lugano, Lugano, Canton Ticino, Switzerland